CLINICAL TRIAL: NCT01592097
Title: A Non-randomized, Exploratory, Study to Assess Clinical Response to Gilenya® (Fingolimod) in a Cohort of Relapsing Remitting Hispanic MS Forms
Brief Title: Exploratory Study to Assess Clinical Response to Gilenya® (Fingolimod) in Hispanics With RRMS
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Lilyana Amezcua, Assistant Professor of Neurology, University of Southern California
Other Study IDs: CFTY720DUS04T
Record Dates: First submitted 2012-05-01; First posted 2012-05-07 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; Autoimmune
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from isolated cells; the remaining cells will be cryopreserved for any duplicate analyses.
Oversight: Data Monitoring Committee: No

SUMMARY:
Gilenya (fingolimod) is approved for multiple sclerosis. However, it is unclear of its clinical effect in the Hispanics with MS given that clinical studies had limited representation of this population. It is also unclear if Gilenya would be as effective in individuals with disease predominantly affecting the optic nerve and spinal cord (OSMS) commonly seen in Asian populations.

Objectives: To compare the clinical response of Gilenya® (fingolimod) in relapsing remitting OSMS and MS of Hispanic descent using ancestral markers as a biomarker of treatment response and clinical disease state.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the success of Gilenya® (fingolimod) treatment in patients with MS of Hispanic descent relative to their ancestral background. Therapeutic success will be determined by annualized relapse rate (ARR; defined as the number of relapses divided by the person years followed) after initiation of treatment with Gilenya® (fingolimod)in comparison to the relapse rate in the previous 12 months. This will be determined based on medical chart extraction, in-person assessment and regular clinical follow-up.

A secondary objective of this study is to investigate whether the efficacy of Gilenya® (fingolimod) is superior or equal in HW which have higher loads of Amerindian versus Caucasian background with opticospinal MS (OSMS-NMO neg) versus classical MS (CMS) in the first 12 months using radiological and clinical parameters. The following measures will be obtained:

1. Number of relapse-free patients over the investigational period
2. Site of relapse defined as brain or spinal cord.
3. Sustained Disability progression will be defined as a one point (1) increase from baseline in patients with baseline EDSS score from 0 to 5.0; or half a point (0.5) increase in patients with baseline EDSS score of 5-5.5 or above after 3 months.
4. MRI changes as described as number of new T2 lesions and number of Gd-enhancing lesions after 12 months from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite multiple sclerosis defined by McDonald Criteria (8) with a score of 0 to 5.5 on the Expanded Disability Status Scale (EDSS)(9). Inclusion will also be determined by PI if clinically indicated. Relapsing remitting form of MS.
* Between 18-65 years of age (This age range is selected so as to capture the vast majority of patients who are seen in the clinics with a confirmed diagnosed of MS. This age range also allows for exclusion of co-morbid conditions that may be associated with aging as well as pediatric cases where their disease characteristics have been shown to be different).
* Ability to understand and sign the IRB-approved informed consent form prior to the performance of any study-specific procedures and is willing to comply with the required scheduling and assessments of the protocol.
* Women of childbearing potential must have a negative urine pregnancy test at the Screening Visit and must be willing to practice a reliable birth-control method.
* Patient must be willing to discontinue and remain free from concomitant immunosuppressive or additional immunomodulatory treatment (including IFNβ1a, 1b, natalizumab and GA) for the duration of the study.
* Willing to answer a series of questions about disease, ancestry, residence history, socioeconomic status and ethnic background.
* Willing to donate 50cc of blood for genetic admixture and immunological testing on three occasions (O months, 6 months, 12 months).
* Willing to undergo MRI as standard of care at a 1.5 Tesla magnet strength at least.

Exclusion Criteria:

* Inability to understand nature of the study.
* Lack of a definite diagnosis of Multiple Sclerosis such as clinical isolated syndrome will be excluded.
* NMO Antibody positive.
* Primary progressive or secondary progressive MS.
* Inability to undergo an MRI study or receive contrast agent and GFR<30.
* Considered by the Investigator to be immunocompromised, based on medical history, physical examination, or laboratory testing or due to prior immunosuppressive treatment.
* Lack of Varicella immunity.
* History of, or available abnormal laboratory results indicative of, any significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric (including major depression), renal, and/or other major disease.
* History of malignancy (subjects with basal cell carcinoma that has been completely excised prior to study entry remain eligible).
* Known history of human immunodeficiency virus infection, hematological malignancy, or organ transplantation, history of severe allergic or anaphylactic reactions or known drug hypersensitivity.
* Prior treatment history with the interferons, glatiramer acetate or natalizumab will be acceptable after drug clearance of 1 month. 1 month has been selected due to clinical experience of possible disease breakthrough if longer period is performed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit 50 individuals with MS who self identify Hispanic descent and are served at USC clinics. Hispanic patients with clinically definite MS, defined by the newly revised McDonald criteria, will be offered the opportunity to participate in this study and asked to give informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2012-06; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lilyana Amezcua, MD, Principal Investigator — University of Southern California
Locations (1):
- Keck School of Medicine of the University of Southern Calfornia, Los Angeles, California, United States

REFERENCES:
- See also: USC MS Comprehensive Care Center and Research Group — https://ms.keckmedicine.org/